CLINICAL TRIAL: NCT06022757
Title: A Phase Ib/II Study of XNW5004 Tablet in Combination With KEYTRUDA® (Pembrolizumab) in Subjects With Advanced Solid Tumors Who Failed Standard Treatments (KEYNOTE F19)
Brief Title: Study of XNW5004 Tablet in Combination With KEYTRUDA® (Pembrolizumab) in Subjects With Advanced Solid Tumors Who Failed Standard Treatments (KEYNOTE F19)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XNW5004-Ib/II-04; KEYNOTE F19 (Other: Merck Sharp & Dohme LLC); MK-3475-F19 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-08-17; First posted 2023-09-05 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma; Squamous Cell Carcinoma of Head and Neck; Urothelial Carcinoma; Prostate Cancer; Small-cell Lung Cancer; Non-small Cell Lung Cancer; Cervical Cancer; Other Solid Tumors
Keywords: XNW5004; EZH2 inhibitor; KEYTRUDA® (pembrolizumab); immune checkpoint inhibitors
MeSH Terms: conditions — Carcinoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell; Prostatic Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms | interventions — pembrolizumab; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Dose escalation and Safety of XNW5004 in combination with KEYTRUDA® (pembrolizumab) (Phase Ib) (Experimental): Dose escalation and safety with repeated administrations of XNW5004 in combination with infusions of KEYTRUDA® (pembrolizumab) in patients with advanced solid tumors.
  Interventions: Drug: XNW5004; Drug: KEYTRUDA® (pembrolizumab) 25 mg/mL Solution for Injection
- HNSCC：XNW5004 in combination with KEYTRUDA® (pembrolizumab) (Phase II - cohort 1) (Experimental): Repeated administrations of XNW5004 in combination with infusions of KEYTRUDA® (pembrolizumab) in patients with head and neck squamous cell carcinoma (including nasopharyngeal carcinoma), urothelial carcinoma, metastatic castration-resistant prostate adenocarcinoma, small cell lung cancer, non-small cell lung cancer, other solid tumor (including cervical cancer)
  Interventions: Drug: XNW5004; Drug: KEYTRUDA® (pembrolizumab) 25 mg/mL Solution for Injection
- Urothelial carcinoma：XNW5004 in combination with KEYTRUDA® (pembrolizumab) (Phase II - cohort 2) (Experimental): Repeated administrations of XNW5004 in combination with infusions of KEYTRUDA® (pembrolizumab) in patients with urothelial carcinoma
  Interventions: Drug: XNW5004; Drug: KEYTRUDA® (pembrolizumab) 25 mg/mL Solution for Injection
- mCRPC：XNW5004 in combination with KEYTRUDA® (pembrolizumab) (Phase II - cohort 3) (Experimental): Repeated administrations of XNW5004 in combination with infusions of KEYTRUDA® (pembrolizumab) in patients with metastatic castration-resistant prostate adenocarcinoma
  Interventions: Drug: XNW5004; Drug: KEYTRUDA® (pembrolizumab) 25 mg/mL Solution for Injection
- Small cell lung cancer：XNW5004 in combination with KEYTRUDA® (pembrolizumab) (Phase II - cohort 4) (Experimental): Repeated administrations of XNW5004 in combination with infusions of KEYTRUDA® (pembrolizumab) in patients with small cell lung cancer
  Interventions: Drug: XNW5004; Drug: KEYTRUDA® (pembrolizumab) 25 mg/mL Solution for Injection
- non-small cell lung cancer:XNW5004 in combination with KEYTRUDA®(pembrolizumab)(PhaseII-cohort5) (Experimental): Repeated administrations of XNW5004 in combination with infusions of KEYTRUDA®(pembrolizumab) in patients with non-small cell long cancer
  Interventions: Drug: XNW5004; Drug: KEYTRUDA® (pembrolizumab) 25 mg/mL Solution for Injection
- ：XNW5004 in combination with KEYTRUDA® (pembrolizumab) (Phase II - cohort 6) (Experimental): Repeated administrations of XNW5004 in combination with infusions of KEYTRUDA® (pembrolizumab) in patients with other solid tumor (including cervical cancer)
  Interventions: Drug: XNW5004; Drug: KEYTRUDA® (pembrolizumab) 25 mg/mL Solution for Injection

INTERVENTIONS:
Drug: XNW5004 — XNW5004 an EZH2 inhibitor, BID, administered in continuous
Drug: KEYTRUDA® (pembrolizumab) 25 mg/mL Solution for Injection — KEYTRUDA® (pembrolizumab) a programmed death receptor (PD-1) blocking antibody administered at 200mg by intravenous (IV) infusions every 3 weeks.

SUMMARY:
In this study, participants with different types of advanced solid tumors who failed standard treatments will be treated with XNW5004 in combination with KEYTRUDA® (pembrolizumab) .

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form prior to the commencement of any research activity/procedure.
* Age ≥ 18.
* Cohort 3 (mCRPC cohort) is male-only, and no gender restrictions for other cohorts.
* Subjects with advanced solid tumors who meet one of the following requirements can be enrolled in the study. No cohorts planned for the Phase Ib study, whereas the Phase II study is divided into 6 cohorts:

  * Cohort: 1 Histologically or cytologically confirmed recurrent or metastatic head and neck squamous cell carcinoma (including nasopharyngeal carcinoma),has progressed after treatment with a standard regimen containing PD-1/PD-L1 inhibitors.
  * Cohort 2: Histologically confirmed advanced urothelial carcinoma (including urothelial carcinoma of bladder, renal pelvis, ureter, and urethral origin) that is not suitable for surgical treatment and has progressed after treatment with a standard regimen containing PD-1/PD-L1 inhibitors.
  * Cohort 3:

    1. Metastatic castration-resistant prostate adenocarcinoma with histological or cytological evidence of disease progression except neuroendocrine or small cell carcinoma; Imaging examination (CT/MRI/ bone scan) confirmed metastatic lesions.
    2. Failed previous standard treatments, and at least received one second-generation anti-androgen drug treatment (including but not limited to abiraterone acetate, enzalutamide or apalutamide).
    3. Disease progression at screening.
    4. Continuous luteinizing hormone-releasing agonist (LHRHa) or antagonist therapy (drug castration) or prior bilateral orchiectomy (surgical castration).
    5. Testosterone at screening was at castration level.
  * Cohort 4: Subjects with histologically or cytologically confirmed extensive-stage small cell lung cancer with disease progression after first-line standard therapy.
  * Cohort 5: Subjects with histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer.

    1. Cohort 5a: Previous use of and resistant to EGFR inhibitors and failed standard treatment.
    2. Cohort 5b: No driver gene mutations identified and failed standard therapy containing PD-1/PD-L1 inhibitors.
  * Cohort 6: Subjects with advanced solid tumors other than those described in the above cohorts, and failed standard therapy. For recurrent or metastatic cervical cancer, it should be histologically or cytologically confirmed as squamous cell carcinoma, progressed after systematic standard treatment, and is not suitable for radical therapy .
* For patients who have progressed on treatment with PD-1/PD-L1 inhibitors administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies, PD-1/PD-L1 inhibitor treatment progression is defined by meeting all of the following criteria:

  1. Has received at least 2 doses of approved PD-1/PD-L1 inhibitors.
  2. Documented objective radiographic progression following initiation of treatment with a PD-1/PD-L1 inhibitor. Subjects should not be enrolled if they are suspected of permanent withdrawal due to pseudo-progression after previous PD-1/PD-L1 inhibitor treatment.
* To the extent possible, provide formalin-fixed, paraffin-embedded (FFPE) tumor tissue section (previously archived or fresh) samples and blood samples that meet the detection requirements for exploratory studies.
* Life expectancy ≥ 3 months.
* At least one measurable lesion according to RECIST 1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Have adequate organ function.
* Females of child-bearing potential and males who use adequate birth control through 6 months post last dose.

Exclusion Criteria:

* Cohort-specific exclusion criteria:

  1. Cohort 1 (head and neck squamous cell carcinoma cohort)

     * Neuroendocrine carcinoma and small cell carcinoma.
     * Salivary adenocarcinoma or other non squamous cell carcinoma (such as adenocarcinoma, sarcoma or mixed carcinoma) confirmed by histology or cytology, and metastatic squamous cell carcinoma with unknown primary origin. This exclusion criterion is not applicable to nasopharyngeal cancer.
  2. Cohort 3 (mCRPC)

     * Severe bone injury caused by tumor bone metastasis, including severe, uncontrolled bone pain as judged by the investigator, bone fractures or spinal cord compression at critical parts of the body that occurred in the last 6 months or are expected to occur in a near future.
     * Any previous treatment targeting T-cell co-stimulation or checkpoint pathways.
  3. Cohort 5 (non-small cell lung cancer)

     * Any previous treatment targeting T-cell co-stimulation or checkpoint pathways other than PD-1 / PD-L1 inhibitors.
     * Combined with other targetable driver mutations either alone or in addition to EGFR, including but not limited to: ALK gene rearrangement, ROS1 mutations, BRAFV600E mutation, etc. (For cohort 5a only.)
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher irAE.
* Prior exposure to EZH2 inhibitor(s) or EZH1/2 inhibitor(s) (including but not limited to tazemetostat).
* Subjects known to be allergic to the study drug or its active ingredients or excipients, or subjects with prior severe hypersensitivity to other monoclonal antibody therapy in the past.
* Subjects who received anti-tumor therapies including chemotherapy, immunotherapy, radical radiotherapy, major surgery, targeting therapy and other anti-tumor therapies within 4 weeks or 5 half-lives of the drug (whichever is shorter) before the first dose; or received palliative radiotherapy within 2 weeks before the first dose.
* Subjects who participated in any other clinical trial of anti-tumor therapy within 28 days before the first dosing, and the last dose of other anti-tumor trial drug is within 28 days prior to the first administration of study drug in this trial.
* Subjects who underwent major surgery within 4 weeks prior to the start of the study treatment, or who are scheduled to undergo a major surgery during the study period (procedures such as puncture or lymph node biopsy is allowed).
* Subjects who have an allogenic bone marrow transplantation or solid organ transplantation.
* Subjects who have diseases requiring systemic therapy with corticosteroids (> 10 mg of prednisone or equivalent dose of other glucocorticoids) or other immunosuppressive medications within 14 days prior to the study drug administration. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal replacement therapy is allowed with a dose of ≤ 10 mg of prednisone or equivalent doses of other glucocorticoids.
* Subjects who took moderate to strong CYP3A4 inhibitor/inducer medications within 14 days prior to the first dose of study drug.
* Subjects who have received live vaccines (including attenuated live vaccines) within 28 days prior to the administration of study drug. Inactivated vaccines are permitted.
* Subjects who experienced toxicity events during previous anti-tumor treatment and the toxicity has not resolved (toxicity has not resolved means the severity of the toxicity events has not been graded as ≤ level 1 according to National Cancer Institute- Common Terminology Criteria for Adverse Events [NCI-CTCAE] 5.0). Other toxicities that the investigator does not think it will affect the safety assessment of the subject (such as hair loss, etc.) will be allowed.
* Subjects who have a history of other malignancies within 3 years prior to enrollment and do not meet the criteria for clinical cure. This exclusion criterion does not apply to skin basal cell carcinoma or squamous cell carcinoma with local treatment methods available and has been cured, superficial bladder cancer, primary cervical carcinoma in situ, intraductal breast carcinoma in situ, and papillary thyroid carcinoma.
* Subjects who have symptoms of active central nervous system metastases. However, subjects with stable brain parenchymal metastases can be enrolled.
* Subjects who have active autoimmune disease that has received systemic treatment in the past 2 years (i.e., taking disease control medications, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered to be systemic treatments.
* Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease. Has had a history of radiation pneumonitis.
* Subjects who have serious psychiatric illness and are unable to cooperate in completing the clinical study.
* Has an active infection requiring systemic therapy.
* Has tuberculosis that is being treated.
* Subjects who have known history of human immunodeficiency virus (HIV) or Anti- Treponema Pallidum test (anti-TP) positive.
* Known acute or chronic active hepatitis B (HBsAg positive or HBcAb positive, and HBV DNA ≥ 200 IU/mL or ≥ 10^3 copies/mL) or acute or chronic active hepatitis C (HCV antibody positive and positive for HCV RNA test).
* Subjects who have history of T-cell lymphoblastic lymphoma (T-LBL) or T-cell lymphoblastic leukemia (T-ALL).
* Subjects who have history of any myeloid malignancies including myelodysplastic syndrome (MDS), or subjects who have abnormal test results related to MDS or myeloproliferative neoplasm (MPN).
* Women during pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of XNW5004 in Combination With KEYTRUDA® (pembrolizumab) (Phase 1b Only) | The first 21-day cycle of therapy
  Recommended Phase 2 dose (RP2D) of XNW5004 as administered orally twice daily (BID), continuously in 21-day cycles, in combination with KEYTRUDA® (pembrolizumab) in subjects with advanced solid tumors by safety data, pharmacokinetic data, pharmacodynamic data and efficacy data
Objective Response Rate (ORR) (Phase 2) | Radiologic tumor assessments performed at baseline(within 28 days before start of study treatment)and every 9 weeks in the first 54 weeks (including the 54th week) after the first drug administration then every 12 weeks thereafter until confirmed disease
  ORR is defined as the proportion of subjects who have a confirmed complete response (CR) or a partial response (PR) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
ORR(Phase 1b) | Radiologic tumor assessments performed at baseline(within 28 days before start of study treatment)and every 9 weeks in the first 54 weeks (including the 54th week) after the first drug administration then every 12 weeks thereafter until confirmed disease
  ORR is defined as the proportion of subjects who have a confirmed CR or a PR per RECIST 1.1.
Duration of response (DOR)(Phase 1b and Phase 2) | Radiologic tumor assessments performed at baseline(within 28 days before start of study treatment)and every 9 weeks in the first 54 weeks (including the 54th week) after the first drug administration then every 12 weeks thereafter until confirmed disease
  DOR is defined defined as the length of time from the date of first confirmed CR or PR per RECIST 1.1(whichever status is recorded first) to the date of first evaluation of progressive disease, or death due to any reasons.
Progression free survival (PFS) (Phase 1b and Phase 2) | Radiologic tumor assessments performed at baseline(within 28 days before start of study treatment)and every 9 weeks in the first 54 weeks (including the 54th week) after the first drug administration then every 12 weeks thereafter until confirmed disease
  PFS is defined as the the length of time from the date of first administration of the study drug until the date of disease progression or death.
Percentage of Participants With Adverse Events（AE） (Phase 2） | Up to 2.5 years
  An AE is any untoward medical occurrence in a clinical investigation subject administered a study drug and an AE can therefore be any symptom, disease or an abnormal laboratory finding, whether or not related to the investigational product. Severity of AEs is assessed according to Common Terminology Criteria for Adverse Events Version (CTCAE 5.0).
Maximum Concentration (Cmax) of XNW5004 in Solid Tumor Participants (Phase 1 and Phase 2） | Cycle 1 (each cycle is 21 days)
  Blood samples were collected at specified intervals for the determination of Cmax.
the area under the plasma concentration-time curve at steady state (AUCss) in Solid Tumor Participants (Phase 1 and Phase 2） | Cycle 1 (each cycle is 21 days)
  Blood samples were collected at specified intervals for the determination of AUCss.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — botanic physician
Locations (1):
- Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, Guodong Province, China

IPD SHARING:
Plan to Share IPD: No